CLINICAL TRIAL: NCT01075802
Title: A Multi-Centre Study of Tamoxifen Dose Escalation Study in Breast Cancer Patients With CYP2D6 Polymorphisms
Brief Title: Study of Tamoxifen Dose Escalation in Breast Cancer Patients With CYP2D6 Polymorphisms
Acronym: TADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Collaborators: St George Hospital, Australia (Other)
Responsible Party: Principal Investigator, Howard Gurney, A/Prof Howard Gurney, Western Sydney Local Health District
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TADE study
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; CYP2D6 Polymorphism
Keywords: Breast cancer; Tamoxifen; Endoxifen; polymorphism of CYP2D6
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamoxifen (Experimental): Dose escalation of tamoxifen in patients with low endoxifen levels
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Dose escalation

SUMMARY:
Tamoxifen is an important drug for the treatment of breast cancer. Used adjuvantly after operation in early breast cancer, tamoxifen reduces annual recurrence rate by half and cancer death by one third. Used preventatively it also reduces the risk of breast cancer by 50% in women at high risk for developing the disease Tamoxifen needs to be activated in the body to an active form called endoxifen, mainly by the enzyme called CYP2D6. Patients have variable capability to activate tamoxifen due to variable function of this enzyme. Studies showed clear correlation of specific genetic variant of CYP2D6 with endoxifen blood levels. It is estimated that up to 25% Caucasian population have reduced or even absent CYP2D6 function. More recently, there were studies that showed the correlation with genetic variant of CYP2D6 and breast cancer relapse in early breast cancer patients treated with tamoxifen. Food and Drug Authority (FDA) in America and recommended checking CYP2D6 genotype in patients receiving tamoxifen treatment, but they did not specify how to interpret the genotype results and what kind actions to take in patient with adverse genotype. The aim of the investigators study is to see if increasing tamoxifen in patients with genetic polymorphism of CYP2D6 will increase endoxifen level to the same range of most patients who have wild type (normal functional)CYP2D6.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status ≤ 1
* Life expectancy ≥ 6 months
* Histologically or cytologically confirmed early, locally advanced or metastatic breast cancer
* Oestrogen receptor positive
* About to start tamoxifen treatment or already on tamoxifen 20mg daily
* Adequate hepatic and renal function

Exclusion Criteria:

* Concurrent chemotherapy or radiotherapy
* Treatment with medications that may alter cytochrome P450 (CYP450)3A4/5 and CYP2D6 activities
* History of thrombosis
* History of non-compliance with previous or current treatment;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effects of genotype of CYP2D on plasma and serum concentration of tamoxifen and its metabolites, with consequent recommendation for dosage adjustment | dose escalation over 40 weeks
To test whether Tamoxifen dose escalation in patients with genetic polymorphism of CYP2D6 will increase endoxifen blood levels to a target level | Dose escalation over 40 weeks
Correlate tamoxifen and its metabolites concentration with tamoxifen side effects | dose escalation over 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard Gurney, MBBS,FRACP, Principal Investigator — South West Sydney Local Health District
Locations (2):
- Australia (2):
  - St George Hospital, Sydney, New South Wales
  - Westmead Cancer Care Centre, Westmead, New South Wales